CLINICAL TRIAL: NCT02127996
Title: A Study to Investigate the Protective Effects of Glucagon-like Peptide-1 (GLP-1) in Patients Undergoing Elective Angioplasty and Stenting (GOLD-PCI)
Brief Title: GLP-1 Loading During Elective Percutaneous Coronary Intervention
Acronym: GOLD-PCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01799
Record Dates: First submitted 2014-04-24; First posted 2014-05-01 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Angina Pectoris; Myocardial Infarction; Reperfusion Injury; Coronary Heart Disease
Keywords: Angina Pectoris; Percutaneous Coronary Intervention; Myocardial Infarction; Glucagon-Like Peptide 1; Reperfusion Injury
MeSH Terms: conditions — Angina Pectoris; Myocardial Infarction; Reperfusion Injury; Coronary Disease | interventions — Glucagon-Like Peptide 1; glucagon-like peptide 1 (7-36)amide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Infusion of Normal Saline during Percutaneous Coronary Intervention
  Interventions: Drug: placebo
- GLP-1 (Experimental): Infusion of GLP-1 (7-36) amide during elective percutaneous coronary intervention
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — GLP-1 (7-36) amide infused at 1.2 pmol/Kg/min
  Other Names: GLP-1 (7-36) amide
  Arms: GLP-1
Drug: placebo — Normal saline
  Arms: Normal Saline

SUMMARY:
Angina is caused by narrowings or blockages within coronary arteries. Coronary angioplasty and stenting is performed for people with angina to improve the blood supply to the heart by placing metal tubes within the artery using balloon inflation. The procedure risks small but significant damage to the heart muscle downstream of the balloon.

Glucagon like peptide 1 (GLP 1) is a naturally occurring hormone secreted by cells in the gut in response to food. It acts by stimulating the release of insulin. In the heart it acts to increase glucose uptake into cardiac muscle. GLP-1 can protect the heart and improve heart muscle performance in people with coronary artery disease in physiological studies. This study which assesses whether GLP-1 protects the heart during coronary angioplasty and stenting.

The hypothesis is that GLP-1 given during elective coronary angioplasty and stenting will reduce cardiac troponin rise (a measure of heart muscle damage) compared to placebo.

ELIGIBILITY:
Inclusion criteria:

* Undergoing elective PCI
* Age over 18
* Able to give informed consent

Exclusion criteria:

* Severe co-morbidity (expected life expectancy < 6 months)
* Nicorandil, glibenclamide, sitagliptin, vildagliptin, saxagliptin, linagliptin, liraglutide, exenatide and insulin use
* Women of child bearing age
* Breast-feeding women
* Myocardial infarction within the previous 3 months
* Baseline elevation of Troponin I before PCI
* Chronic Renal Impairment (serum creatinine > 160 μmol/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03-31 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Plasma Troponin I level | 6 Hours following angioplasty or stenting
  Incidence of Troponin I elevation of > 5 x 99th percentile upper reference limit on blood test at approximately 6 hours post procedure.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular or Cerebrovascular Event (MACCE) Rates | From date of randomisation until the date of first event assessed up to 6 months
  MACCE rate (death, stent thrombosis, myocardial infarction, acute coronary syndrome, hospitalisation with heart failure, stroke)- these will be patient reported and confirmed by interrogation of hospital records and interrogation of local and national databases.
Plasma Creatine Kinase - Myocardial Bound (CKMB) level | 6 hours
  CKMB level on blood test at 6 hours following angioplasty or stenting
Myocardial Flow Grade after Angioplasty or Stenting | Measured during procedure
  Graded between 0 and 3 on Thrombolysis in Myocardial Infarction (TIMI) Scale
MACCE Rates | From date of randomisation until the date of first event assessed up to 12 months
  MACCE rate (death, stent thrombosis, myocardial infarction, acute coronary syndrome, hospitalisation with heart failure, stroke)- these will be patient reported and confirmed by interrogation of hospital records and interrogation of local and national databases.
MACCE Rates | From date of randomisation until the date of first event assessed up to 60 months
  MACCE rate (death, stent thrombosis, myocardial infarction, acute coronary syndrome, hospitalisation with heart failure, stroke)- these will be patient reported and confirmed by interrogation of hospital records and interrogation of local and national databases.
Ischaemic symptoms during balloon occlusion | Assessed during procedure
  Presence or absence or of symptoms of myocardial ischaemia during the procedure
Myocardial Blush Grade following angioplasty or stenting | Measured during procedure
  Graded between 0 and 3 on Thrombolysis in Myocardial Infarction (TIMI) Scale
Electrocardiographic (ECG) Changes during procedure | Assessed during procedure
  Presence or absence of ECG changes reflective of myocardial ischaemia during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hoole, MA MD FRCP, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Giblett JP, Clarke S, Zhao T, McCormick LM, Braganza DM, Densem CG, O'Sullivan M, Adlam D, Clarke SC, Steele J, Fielding S, West NEJ, Villar SS, Hoole SP. The role of Glucagon-Like Peptide 1 Loading on periprocedural myocardial infarction During elective PCI (GOLD-PCI study): A randomized, placebo-controlled trial. Am Heart J. 2019 Sep;215:41-51. doi: 10.1016/j.ahj.2019.05.013. Epub 2019 Jun 9. PMID 31277053